CLINICAL TRIAL: NCT04303663
Title: Randomised Controlled Trial to Compare the Efficacy of Fibular Nail Fixation vs Plate Fixation in Ankle Fracture Management
Brief Title: Fibular Nail vs Plate in Ankle Fractures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Samuel KK Ling, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUHK_fibularnail
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Ankle Fractures
Keywords: Fibular Nail; Fibular Rod; Fibular Plate
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibular Plate (Active Comparator): Open reduction and internal fixation of the fibular fracture Fixation of the fibular will be performed with a fibular plate +/- lag screws as judged intraoperatively
  Interventions: Procedure: Fibular Plate
- Fibular Nail (Experimental): Percutaneous or mini-open reduction of the fibular fracture and fixation with a fibular nail.
  Interventions: Procedure: Fibular Nail

INTERVENTIONS:
Procedure: Fibular Plate — ORIF with Plating
  Arms: Fibular Plate
Procedure: Fibular Nail — CRIF +/- ORIF with Fibular nail
  Arms: Fibular Nail

SUMMARY:
Randomised Controlled Trial to Compare the Efficacy of Fibular Nail Fixation vs Plate Fixation in Ankle Fracture Management

DETAILED DESCRIPTION:
Ankle fracture is a common injury with a wide spectrum of mechanism, especially in the elderly population. Surgical treatment of the unstable ankle fracture presents encouraging outcomes. Open reduction with plate osteosynthesis is the gold standard but is sometimes complicated by wound problems. The overall rate of complications after open reduction and internal fixation of ankle fracture varies from 5% to 40%. Wound complication, including superficial and deep ones, was reported as high as 18.8% in a previous meta-analysis, especially in the patients with high-risk factors e.g. elderly, osteoarthritis and diabetic subpopulation.

Newer implants such as locked fibular nail (FN) have been developed with studies showing promising results. The Acumed fibular rod system is such an alternative method which is a metallic implant with length 110mm, 145 mm and 180 mm. The shorter diameter of the nail (ranging from 3.0 mm-3.6 mm) allows surgeons to make an incision as short as 1 cm compared to the 8-cm incision in conventional lateral plate fixation. Also, it shows advantages in mechanical stability for osteoporotic bone with less prominent metalwork. The nail is anchored by a lateral-medial locking screw at the level of the syndesmosis and two anterior-posterior locking screws distally. A 1-cm longitudinal incision will be made over the tip of the lateral malleolus after performing a closed reduction.

The results from previous studies imply that the fibular rod system may give positive outcomes. However, the majority of the relative studies were single-centre series providing a low level of evidence and lacking a comparative group. For example, a case series retrospectively reviewed 105 patients who experienced surgical treatment using the Acumed fibular rod system for ankle fracture and found good functional and radiographic results with minimal complications. Like all other retrospective studies, the follow up was not complete and some radiographic information could not be obtained. Thus a comparative study with a high level of evidence is required to provide more information for surgeons.

To the investigators' best knowledge, no prospective randomized controlled trials have been conducted to investigate the clinical outcomes and radiographic results after surgical treatment using the Acumed fibular rod system in ankle fracture. The objective of the study is to compare the clinical outcomes of locking fibular nail and to results of the open-reduction with plate fixation in ankle fracture management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with minimally displaced fibular fracture
* Type A or type B according to Weber ankle fracture classification
* Be able to walk without assistance in pre-injury status

Exclusion Criteria:

* Medical co-morbidity that prevents the patient from undergoing surgery
* Surgery delayed for >2-weeks after the initial injury
* Pre-existing/old injury in the ipsilateral limb
* Severe physical, mental disability that renders the participant unable to conform to usual rehabilitation regimes (Recent lower limb surgery, pre-existing neurological problem and etc.)
* Incapable to understand the study protocol or provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Foot Function | 12-week
  Foot and Ankle Outcome Score split into 5 categories: symptoms, pain, ADL, recreation, QOL. 0-100 with 0=severe symptoms and 100=no symptoms.
Foot Function | 26-week
  Foot and Ankle Outcome Score split into 5 categories: symptoms, pain, ADL, recreation, QOL. 0-100 with 0=severe symptoms and 100=no symptoms.

SECONDARY OUTCOMES:
Routine radiological parameters | 0 week
  Standard ankle X-Ray from the anterior-posterior (AP) and lateral projection will be taken. medial and tibiotalar clear space and the talocrural angle will be measured.
Routine radiological parameters | 6-weeks
  Standard ankle X-Ray from the anterior-posterior (AP) and lateral projection will be taken. medial and tibiotalar clear space and the talocrural angle will be measured.
Routine radiological parameters | 12-weeks
  Standard ankle X-Ray from the anterior-posterior (AP) and lateral projection will be taken. medial and tibiotalar clear space and the talocrural angle will be measured.
Routine radiological parameters | 26-weeks
  Standard ankle X-Ray from the anterior-posterior (AP) and lateral projection will be taken. medial and tibiotalar clear space and the talocrural angle will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel KK Ling, MBChB, Principal Investigator — CUHK

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salai M, Dudkiewicz I, Novikov I, Amit Y, Chechick A. The epidemic of ankle fractures in the elderly--is surgical treatment warranted? Arch Orthop Trauma Surg. 2000;120(9):511-3. doi: 10.1007/s004020000172. PMID 11011670
- [Background] Pagliaro AJ, Michelson JD, Mizel MS. Results of operative fixation of unstable ankle fractures in geriatric patients. Foot Ankle Int. 2001 May;22(5):399-402. doi: 10.1177/107110070102200507. PMID 11428758
- [Background] Appleton P, McQueen M, Court-Brown C. The Fibula Nail for Treatment of Ankle Fractures in Elderly and High Risk Patients. Tech Foot Ankle Surg [Internet]. 2006;5(3).
- [Background] Bugler KE, Watson CD, Hardie AR, Appleton P, McQueen MM, Court-Brown CM, White TO. The treatment of unstable fractures of the ankle using the Acumed fibular nail: development of a technique. J Bone Joint Surg Br. 2012 Aug;94(8):1107-12. doi: 10.1302/0301-620X.94B8.28620. PMID 22844054